CLINICAL TRIAL: NCT05263817
Title: A Clinical Study on the Safety and Effectiveness of CD19/BCMA Chimeric Antigen Receptor T Cells in the Treatment of Refractory POEMS Syndrome, Amyloidosis, Autoimmune Hemolytic Anemia, and Vasculitis
Brief Title: A Clinical Study of CD19/BCMA CAR-T Cells in the Treatment of Refractory POEMS Syndrome, Amyloidosis, Autoimmune Hemolytic Anemia, and Vasculitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19/BCMA-005
Record Dates: First submitted 2021-12-01; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: POEMS Syndrome; Amyloidosis; Autoimmune Hemolytic Anemia; Vasculitis
Keywords: CD19 CAR-T; BCMA CAR-T; POEMS Syndrome; Amyloidosis; Autoimmune Hemolytic Anemia; Vasculitis
MeSH Terms: conditions — POEMS Syndrome; Amyloidosis; Anemia, Hemolytic, Autoimmune; Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- POEMS Syndrome (Experimental)
  Interventions: Biological: CD19/BCMA CAR T-cells
- Amyloidosis (Experimental)
  Interventions: Biological: CD19/BCMA CAR T-cells
- Autoimmune Hemolytic Anemia (Experimental)
  Interventions: Biological: CD19/BCMA CAR T-cells
- Vasculitis (Experimental)
  Interventions: Biological: CD19/BCMA CAR T-cells

INTERVENTIONS:
Biological: CD19/BCMA CAR T-cells — Each subject receive CD19/BCMA CAR T-cells by intravenous infusion
  Other Names: CD19/BCMA CAR T-cells injection

SUMMARY:
A Clinical Study on the Safety and Effectiveness of CD19/BCMA Chimeric Antigen Receptor T Cells in the Treatment of Refractory POEMS Syndrome, Amyloidosis, Autoimmune Hemolytic Anemia, and Vasculitis

DETAILED DESCRIPTION:
POEMS syndrome, amyloidosis, autoimmune hemolytic anemia, vasculitis and other diseases may only show local pathological damage or systemic lesions. If they are not diagnosed and treated in time or poorly controlled, they will progress as the course of the disease progresses. Risk of disability or even death.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with POEMS syndrome, amyloidosis, autoimmune hemolytic anemia, vasculitis, and the curative effect of conventional hormones, radiotherapy and chemotherapy, protease inhibitors is not good and (or) no effective treatment means.

  2. After glucocorticoids, cyclophosphamide or methotrexate treatments there are still relapsed and refractory diseases, or clearly show intolerance/toxicity to these drugs.

  3. Estimated survival time> 12 weeks; 4. Patients had a negative urine pregnancy test before the start of administration and agreed to take effective contraceptive measures during the test period until the last follow-up; 5. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* Subjects with any of the following exclusion criteria were not eligible for this trial:

  1. History of craniocerebral trauma, conscious disturbance, epilepsy,cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
  2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythm ia in the past;
  3. Pregnant (or lactating) women;
  4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
  5. Active infection of hepatitis B virus or hepatitis C virus;
  6. Systemic steroids have used in the 4 weeks before participating in the treatment (except recently or currently using inhaled steroids);
  7. Those who have used any gene therapy products before.
  8. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
  9. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
  10. Those who suffer from other uncontrolled diseases are not suitable to join the study;
  11. HIV infection;
  12. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD19/BCMA targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CD19/BCMA targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Titer of auto-antibody Titer of auto-antibody titer of auto-antibody | Up to 2 years after CD19/BCMA targeted CAR T-cells infusion
  In peripheral blood and bone marrow
Overall response rate (ORR) | Up to 2 years after CD19/BCMA targeted CAR T-cells infusion
  Proportion of subjects with complete or partial remission
Best overall response, BOR | At ≤3 month
  Assessment of ORR at ≤3 month
Overall survival (OS) | From CD19/BCMA CAR-T infusion to death，up to 2 years
  The time from the cell reinfusion to death due to any cause
Duration of remission, DOR | 2 years post CD19/BCMA CAR-T cells infusion
  The time from the first assessment of remission or partial remission of the disease to the first assessment of disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China